CLINICAL TRIAL: NCT03547063
Title: Responses to Appetite and Taste in the Brain Circuits That Control Eating Behaviour: An fMRI Study Evaluating Brain Structure, Connectivity and Responses to Taste Across Different Body Weight Categories and in Response to Weight Loss
Brief Title: Responses to Appetite and Taste in the Brain Circuits That Control Eating Behaviour
Acronym: TASTER
Status: Suspended | Type: Observational
Why Stopped: COVID-19
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 18/0233
Record Dates: First submitted 2018-05-11; First posted 2018-06-06 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Obesity
Keywords: Obesity, appetite, taste, fMRI
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, plasma and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sleeve Gastrectomy (SG): 25 participants, male and female, aged 18-50 years, body mass index (BMI) 35-50 kg/m2, due to undergo primary SG
- Lifestyle Intervention: 25 participants, male and female, aged 18-50 years, BMI 35-50 kg/m2
- Normal Weight: 25 participants, aged 18-50 years BMI 18.5-24.9 kg/m2, age and gender matched to group with severe obesity

SUMMARY:
The aim of this study is to gain insight into brain structure and the neural networks that control taste and eating behaviour in patients with severe obesity undergoing a primary sleeve gastrectomy (SG) or a lifestyle intervention for weight loss compared with normal weight individuals, using functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
This is an observational study aiming to gain insight into brain structure and the neural networks that control taste and eating behaviour in patients with severe obesity undergoing a primary sleeve gastrectomy (SG) or a lifestyle intervention for weight loss compared with normal weight individuals using functional magnetic resonance imaging (fMRI). Drops of liquid foods and a control solution will be delivered to the participants' mouth during fMRI scanning. Body weight, gut hormones from serial blood samples, appetite scores and taste will be assessed at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Female and male adults aged 18-50 years.
* Right-handed.
* No MRI contra-indications.
* Weight stable at time of recruitment, defined as less than 5% variation in body weight over the preceding 3 months.
* Proficient in written and spoken English.
* Able to comply with study protocol.
* Willing and able to provide written informed consent.
* Participants must be registered with a general practitioner (GP).
* Willing for their treating consultant or their GP and the study team to be informed in the event of an incidental abnormal finding being detected by the investigations or assessments that form part of this study.
* Able to lie flat for 1 hour.

Group-specific inclusion criteria:

* SG group:

  * BMI of 35-50 kg/m2
  * Planned to undergo primary SG surgery and fulfilling eligibility criteria for bariatric surgery.
* Lifestyle intervention group:

  * BMI of 35-50 kg/m2
  * Willing to undergo a lifestyle intervention programme with a view to achieving approximately 10% weight loss.
* Normal weight group:

  * BMI 18.5-24.9 kg/m2

Exclusion Criteria:

* Body weight greater than 130kg (due to weight limit of MRI Scanner).
* Contraindications specific to MRI scanning: metallic implants (cardiac pacemakers, aneurysm clips, permanent eye lining, cochlear implants or anyone who has been exposed to metallic flakes or splinters).
* Type 1 and type 2 diabetes (in view of altered circulated gut hormone profiles and gustatory function).
* Menopause (in view of findings that the menopause affects gustatory function).
* Smoking (in view of the fact that smoking affects salivary gut hormones and gustatory function).
* Vitamin B12 or zinc deficiency (in view of deficiencies affecting gustatory function).
* Untreated severe depression.
* Eating disorders including bulimia and self-induced vomiting.
* Neurological or psychiatric conditions.
* Acute illness or chronic conditions that may impact upon gustatory and olfactory function.
* Acute illness or chronic conditions that may impact upon post-operative weight loss.
* Known or suspected history of HIV, Hepatitis B or C or other blood-borne diseases (in view of safety regulations regarding exposure to blood products)
* Pregnancy or lactation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participant groups:
  1. Participants with severe obesity
     1. SG: 25 participants, male and female, aged 18-50 years, body mass index (BMI) 35-50 kg/m2, due to undergo primary SG.
     2. Lifestyle intervention: 25 participants, male and female, aged 18-50 years, BMI 35-50 kg/m2.
  2. Participants with normal weight: 25 participants, aged 18-50 years BMI 18.5-24.9 kg/m2, age and gender matched to group with severe obesity.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2018-12-18 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
BOLD signal change after SG | approximately 6 weeks
  To determine the effect of SG, at 10% weight loss, upon whole-brain neural response to taste, in the fed and fasted state, detected through blood-oxygen-level dependent (BOLD) signal, in patients with severe obesity.

SECONDARY OUTCOMES:
BOLD signal change after lifestyle intervention | average of 12 weeks
  The effect of 10% weight loss in patients with severe obesity induced by a lifestyle intervention on BOLD signal to taste in the fed and fasted state and compared to SG.
BOLD signal in response to taste in severe obesity compared to normal weight | baseline
  Brain responses, as BOLD signal, to taste in the fed and fasted state in severe obesity compared to normal weight
BOLD signal change post-SG | 6 months
  Whole brain neural response in BOLD signal to taste, in the fed and fasted state, 6 months following SG versus normal weight
Correlation of taste responses and gut hormones | baseline
  The relationship between the neural correlates of taste and levels of circulating gut hormones in severe obesity compared to normal weight
Correlation of taste responses and gut hormones | approximately 6 weeks for SG group and approximately 12 weeks for lifestyle intervention group
  The relationship between the neural correlates of taste and levels of circulating gut hormones after 10% weight loss by SG compared to lifestyle intervention
Correlation of taste responses and gut hormones | 6 months post-SG compared to baseline
  The relationship between the neural correlates of taste and circulating gut hormone levels
Correlation of taste responses and gut hormones | 6 months
  The relationship between the neural correlates of taste and levels of circulating gut hormones post-SG compared to normal weight
Brain structure | Baseline
  Comparison of brain structure in severe obesity and normal weight
Brain structure 6 months following SG | 6 months
  Comparison of brain structure 6 months following SG to baseline
Brain structure after 10% weight loss | approximately 6 weeks for SG group and approximately 12 weeks for lifestyle intervention group
  Comparison of brain structure following 10% weight loss induced by SG versus lifestyle intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Batterham, PhD FRCP, Principal Investigator — UCL
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Makaronidis JM, Neilson S, Cheung WH, Tymoszuk U, Pucci A, Finer N, Doyle J, Hashemi M, Elkalaawy M, Adamo M, Jenkinson A, Batterham RL. Reported appetite, taste and smell changes following Roux-en-Y gastric bypass and sleeve gastrectomy: Effect of gender, type 2 diabetes and relationship to post-operative weight loss. Appetite. 2016 Dec 1;107:93-105. doi: 10.1016/j.appet.2016.07.029. Epub 2016 Jul 22. PMID 27453553
- [Background] Batterham RL, ffytche DH, Rosenthal JM, Zelaya FO, Barker GJ, Withers DJ, Williams SC. PYY modulation of cortical and hypothalamic brain areas predicts feeding behaviour in humans. Nature. 2007 Nov 1;450(7166):106-9. doi: 10.1038/nature06212. Epub 2007 Oct 14. PMID 17934448
- [Background] Neseliler S, Han JE, Dagher A. The Use of Functional Magnetic Resonance Imaging in the Study of Appetite and Obesity. In: Harris RBS, editor. Appetite and Food Intake: Central Control. 2nd edition. Boca Raton (FL): CRC Press/Taylor & Francis; 2017. Chapter 6. Available from http://www.ncbi.nlm.nih.gov/books/NBK453146/ PMID 28880516
- [Background] Zhang Y, Ji G, Xu M, Cai W, Zhu Q, Qian L, Zhang YE, Yuan K, Liu J, Li Q, Cui G, Wang H, Zhao Q, Wu K, Fan D, Gold MS, Tian J, Tomasi D, Liu Y, Nie Y, Wang GJ. Recovery of brain structural abnormalities in morbidly obese patients after bariatric surgery. Int J Obes (Lond). 2016 Oct;40(10):1558-1565. doi: 10.1038/ijo.2016.98. Epub 2016 May 20. PMID 27200505
- [Background] Goldstone AP, Miras AD, Scholtz S, Jackson S, Neff KJ, Penicaud L, Geoghegan J, Chhina N, Durighel G, Bell JD, Meillon S, le Roux CW. Link Between Increased Satiety Gut Hormones and Reduced Food Reward After Gastric Bypass Surgery for Obesity. J Clin Endocrinol Metab. 2016 Feb;101(2):599-609. doi: 10.1210/jc.2015-2665. Epub 2015 Nov 18. PMID 26580235
- [Background] Faulconbridge LF, Ruparel K, Loughead J, Allison KC, Hesson LA, Fabricatore AN, Rochette A, Ritter S, Hopson RD, Sarwer DB, Williams NN, Geliebter A, Gur RC, Wadden TA. Changes in neural responsivity to highly palatable foods following roux-en-Y gastric bypass, sleeve gastrectomy, or weight stability: An fMRI study. Obesity (Silver Spring). 2016 May;24(5):1054-60. doi: 10.1002/oby.21464. PMID 27112067
- [Background] Karra E, O'Daly OG, Choudhury AI, Yousseif A, Millership S, Neary MT, Scott WR, Chandarana K, Manning S, Hess ME, Iwakura H, Akamizu T, Millet Q, Gelegen C, Drew ME, Rahman S, Emmanuel JJ, Williams SC, Ruther UU, Bruning JC, Withers DJ, Zelaya FO, Batterham RL. A link between FTO, ghrelin, and impaired brain food-cue responsivity. J Clin Invest. 2013 Aug;123(8):3539-51. doi: 10.1172/JCI44403. Epub 2013 Jul 15. PMID 23867619